CLINICAL TRIAL: NCT01610635
Title: A Randomised Trial to Determine Whether the Interval Between Blood Donations in England Can be Safely and Acceptably Decreased
Brief Title: INTERVAL Study: To Determine Whether the Interval Between Blood Donations in England Can be Safely and Acceptably Decreased
Acronym: INTERVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cambridge (Other)
Collaborators: National Health Service, Blood and Transplant (Unknown); University of Oxford (Other)
Responsible Party: Principal Investigator, Professor Danesh, Professor of Epidemiology and Medicine, Head of Department of Public Health and Primary Care, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-01-GEN; 24760606 (Other: ISRCTN)
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Blood Donation
Keywords: RCT; blood donation frequency; quality of life; iron deficiency
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Male - 8 weeks (Experimental): Male donors assigned to an 8 week donation interval frequency
  Interventions: Other: Reduced versus standard intervals between blood donations
- Male - 10 weeks (Experimental): Male donors assigned to 10 week donation interval frequency
  Interventions: Other: Reduced versus standard intervals between blood donations
- Male - 12 weeks (No Intervention): Male donors assigned to 12 week donation interval frequency
- Female - 12 weeks (Experimental): Female donors assigned to 12 week donation interval frequency
  Interventions: Other: Reduced versus standard intervals between blood donations
- Female - 14 weeks (Experimental): Female donors assigned to 14 week donation interval frequency
  Interventions: Other: Reduced versus standard intervals between blood donations
- Female - 16 weeks (No Intervention): Female donors assigned to 16 week donation interval frequency

INTERVENTIONS:
Other: Reduced versus standard intervals between blood donations — Over a period of two years participants will be invited to give blood either at usual donation intervals or more frequently. Men will be invited to donate every 12, 10 or 8 weeks and women every 16, 14 or 12 weeks.
  Arms: Female - 12 weeks; Female - 14 weeks; Male - 10 weeks; Male - 8 weeks

SUMMARY:
It is hypothesised that the number of donations made by English blood donors will be greater with reduced vs. standard inter-donation intervals. The null hypothesis is that there will be no difference in donations between treatment groups; this may arise if reduced inter-donation intervals result in a greater number of donation deferrals (due to low haemoglobin) and/or an unacceptable burden to donors.

DETAILED DESCRIPTION:
50,000 blood donors will be recruited from permanent blood donation centres across England to compare different intervals between blood donations to try to find the optimum interval for which it is safe for different donors to give blood. The study will look at whether intervals should be tailored by age, gender, genetic profile, and other characteristics. Study findings should help to improve the well-being of future blood donors in England and enhance the country's blood supplies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and fulfilling all normal criteria for blood donation
2. Willing to be assigned to any of the study intervention groups
3. Registered at one of the permanent donation clinics at the time of enrolment

Exclusion Criteria:

* As the aim of the study is to be almost "paper-less", it will involve remote web-based data collection. Hence, participants who do not have internet access and/or are not willing to provide an email address for study correspondence will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Total blood collected after two years | 24 months
  Expressed in units (470ml) per person per year

SECONDARY OUTCOMES:
Donor quality of life | 24 months
  Measured using the SF-36 health survey
Number of donation deferrals | 24 months
  Temporary rejection of donors due to low haemoglobin and other factors
Markers of iron status | 24 months
  Serum ferritin and reticulocyte haemoglobin
Cognitive ability | 24 months
  Reasoning, attention and memory
Levels of physical activity | 24 months
Cost effectiveness | 24 months
Donor attitudes, beliefs and values | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: John Danesh, Principal Investigator — University of Cambridge; David Roberts, Principal Investigator — University of Oxford
Locations (25):
- United Kingdom (25):
  - Brentwood Blood Donor Centre, Brentwood, Essex
  - Edgware Blood Donor Centre, Edgware, Middlesex
  - Birmingham Blood Donor Centre, Birmingham
  - Bradford Blood Donor Centre, Bradford
  - Bristol Blood Donor Centre, Bristol
  - Cambridge Blood Donor Centre, Cambridge
  - Gloucester Blood Donor Centre, Gloucester
  - Lancaster Blood Donor Centre, Lancaster
  - Leeds City Centre Blood Donor Centre, Leeds
  - Leeds Blood Donor Centre, Leeds
  - Leicester Blood Donor Centre, Leicester
  - Liverpool Blood Donor Centre, Liverpool
  - Tooting Blood Donor Centre, London
  - West End Blood Donor Centre, London
  - Luton Blood Donor Centre, Luton
  - Manchester Plymouth Grove, Manchester
  - Manchester Norfolk House Blood Donor Centre, Manchester
  - Newcastle Blood Donor Centre, Newcastle
  - Nottingham Blood Donor Centre, Nottingham
  - Oxford Blood Donor Centre, Oxford
  - Plymouth Blood Donor Centre, Plymouth
  - Poole Blood Donor Centre, Poole
  - Sheffield Blood Donor Centre, Sheffield
  - Southampton Blood Donor Centre, Southampton
  - Stoke Blood Donor Centre, Stoke

REFERENCES:
- See also: ISRCTN study record — http://www.controlled-trials.com/ISRCTN24760606/ISRCTN24760606
- See also: INTERVAL study webpage — http://www.intervalstudy.org.uk